CLINICAL TRIAL: NCT06214273
Title: Evaluation of Low Level Diode Diode Versus Topical Chamomile in Management of Chemotherapy Induced Oral Mucositis: Three Arm Randomized Clinical Trial
Brief Title: Low Level Diode Laser Versus Topical Chamomile in Management of Chemotherapy Induced Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Clair Sobhy Nagieb Botros, Oral medicine specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27283522022441
Record Dates: First submitted 2023-12-13; First posted 2024-01-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Chemotherapy Induced Oral Mucositis
MeSH Terms: interventions — Low-Level Light Therapy; Chamomile extract

STUDY DESIGN:
Intervention Model Description: a three-arm head-to-head RCT assessing two of the promising studied interventions, low-level diode laser and topical chamomile, comparing them to each other's and to conventional therapy.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Double-blinded trial:
  The outcome assessor and the statistician will be blinded. Participants can't be blinded because of the difference in intervention methods of application.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen oral gel and miconazole oral gel (Active Comparator): One group will receive conventional oral therapy composed of topical ibuprofen oral gel as an anti-inflammatory and analgesic and topical miconazole as an anti-fungal oral gel.
  Interventions: Drug: Ibuprofen analgesic and anti-inflammatory oral gel and miconazole anti fungal oral gel
- low-level diode laser diode laser (Experimental): The second group will receive a diode laser with a wave length range of 800-980 nm and power less than 500 ml.
  Interventions: Device: Low level diode laser
- Chamomile (Experimental): The third group will receive chamomile 3% mucoadhesive gel.
  Interventions: Drug: Chamomile

INTERVENTIONS:
Device: Low level diode laser — diode laser with a wave length range of 800-980 n m and power less than 500 ml
  Other Names: Photobiomodulation
  Arms: low-level diode laser diode laser
Drug: Chamomile — Chamomile 3% mucoadhesive gel
  Other Names: Matricaria
  Arms: Chamomile
Drug: Ibuprofen analgesic and anti-inflammatory oral gel and miconazole anti fungal oral gel — Topical anti-inflammatory, topical analgesic and topical antifungal
  Other Names: conventional oral therapy; Ibuprofen oral gel and miconazole oral gel
  Arms: Ibuprofen oral gel and miconazole oral gel

SUMMARY:
a three-arm head-to-head randomized clinical trial assessing two of the promising studied interventions, low-level diode laser and topical Chamomile, comparing them to each other's and to conventional therapy in the management of oral mucositis-induced chemotherapy.

DETAILED DESCRIPTION:
The latest MASCC/ISOO Mucositis Guidelines recommend relieving pain, reducing inflammation, and preventing secondary infection as the main pillars in the management of chemotherapy-induced oral mucositis. Accordingly, our comparator will be conventional therapy, including topical anti-inflammatory, topical analgesic, and topical antifungal.

ELIGIBILITY:
Inclusion criteria:

* Patients with chemotherapy-induced oral mucositis.
* Patients who will agree to participate in the study.
* Adult Patients above 18 years.

Exclusion criteria:

* Patients with any visible oral lesions other than oral mucositis.
* Patients who have received radiotherapy 2 weeks earlier to the diagnosis of the oral mucositis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Discomfort and pain | On baseline, first, third, fifth, seventh, tenth and 14th day.
  Reported by each patient using the Visual Analog Scale (0-10),10 refers to maximum pain

SECONDARY OUTCOMES:
Oral mucositis severity | On baseline, first, third, fifth, seventh, tenth and 14th day.
  It will be measured using the WHO grading Scale (0-4).4 refers to ulcers, and diet is not possible (due to mucositis).
The total healing time of oral ulcers | On baseline, first, third, fifth, seventh, tenth and 14th day.
  will be recorded for all the patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paice JA, Cohen FL. Validity of a verbally administered numeric rating scale to measure cancer pain intensity. Cancer Nurs. 1997 Apr;20(2):88-93. doi: 10.1097/00002820-199704000-00002. PMID 9145556
- [Result] Soares ADS, Wanzeler AMV, Cavalcante GHS, Barros EMDS, Carneiro RCM, Tuji FM. Therapeutic effects of andiroba (Carapa guianensis Aubl) oil, compared to low power laser, on oral mucositis in children underwent chemotherapy: A clinical study. J Ethnopharmacol. 2021 Jan 10;264:113365. doi: 10.1016/j.jep.2020.113365. Epub 2020 Sep 10. PMID 32920135
- [Result] Elhadad MA, El-Negoumy E, Taalab MR, Ibrahim RS, Elsaka RO. The effect of topical chamomile in the prevention of chemotherapy-induced oral mucositis: A randomized clinical trial. Oral Dis. 2022 Jan;28(1):164-172. doi: 10.1111/odi.13749. Epub 2020 Dec 19. PMID 33290635
- [Result] de Lima VHS, de Oliveira-Neto OB, da Hora Sales PH, da Silva Torres T, de Lima FJC. Effectiveness of low-level laser therapy for oral mucositis prevention in patients undergoing chemoradiotherapy for the treatment of head and neck cancer: A systematic review and meta-analysis. Oral Oncol. 2020 Mar;102:104524. doi: 10.1016/j.oraloncology.2019.104524. Epub 2020 Feb 13. PMID 32062592